CLINICAL TRIAL: NCT00449982
Title: A Randomized, Double-Blind, Three-Arm Parallel-Group, Placebo-Controlled Phase 3 Trial to Investigate the Clinical Efficacy and Safety of Polyphenon E in the Treatment of External Genital Warts
Brief Title: Efficacy and Safety Study of Polyphenon E to Treat External Genital Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediGene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT 1018
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Condylomata Acuminata
Keywords: Genital warts; Condylomata acuminata; Human Papillomavirus; Polyphenon E; Green tea extract; Vulva; Penis; Anus
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Polyphenon E Ointment 10%, Polyphenon E Ointment 15%

SUMMARY:
The purpose of this study is to investigate the clinical efficacy, safety and tolerability of a Polyphenon E Ointment 10% and a Polyphenon E Ointment 15% in the treatment of external genitial warts in male and female patients.

DETAILED DESCRIPTION:
External genital warts are non-malignant tumors caused by infections of the human papillomavirus (HPV), mainly types 6 and 11. Genital wart infections have one of the fastest growing incidence rates of all sexually transmitted diseases, with about 1% of sexually active adults in the United States suffering from this infection and at least 15% with subclinical infection. None of the current treatment options (with exception of interferon) has been subjected to controlled prospective clinical trials, although they are generally regarded as safe and effective. However, one of their major disadvantages is that they are painful and may cause scarring. Additionally recurrence of warts can often be observed. Against this background the study tries to evaluate another effective and well tolerated therapeutic option by using an extract of green tea leaves.

Comparison: Polyphenon E Ointment 10%, Polyphenon E Ointment 15%, placebo

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of enrollment
* Clinical diagnosis of external genital warts (located genital, inguinal, perineal or perianal)
* At least 2, but no more than 30 external genital warts
* A total wart area between 12 and 600mm²
* Negative pregnancy test and willingness to use effective contraception (for women of child-bearing potential)
* For partners of male patients who are of child-bearing potential: use of effective contraception during the treatment period
* Written informed consent
* Ability to comply with the requirements of the study

Exclusion Criteria:

* Participation in an investigational trail within 30 days prior to enrollment
* Previous participation in a trial investigating Polyphenon E in the treatment of external genital warts
* Treatment of external genital warts within 30 days prior to enrollment and for the whole study duration
* Systemic intake of virostatics within 30 days prior to enrollment and for the whole study duration
* Systemic intake of immunosuppressive or immunomodulatory medication within 30 days prior to enrollment and for the whole study duration
* Current infection with Herpes genitalis or history of Herpes genitalis infection within the last 3 month
* Any current and/or recurrent pathologically relevant genital infections other than genital warts
* Current known acute or chronic infection with HBV or HCV
* Known HIV infection
* Any current uncontrolled infection
* Organ allograft
* For female patients: pregnancy or lactation
* Known allergies against any of the ingredients of the treatments
* Any chronic or acute skin condition susceptible of interfering with the evaluation of the drug effect
* Any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study
* Internal (vaginal or rectal) warts requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2003-07; Study Completion 2004-08

PRIMARY OUTCOMES:
Complete clearance of all warts within a maximum of 16 weeks treatment
Severe local reaction during the treatment period

SECONDARY OUTCOMES:
Time to complete clearance of all warts, of all baseline warts, and of all new warts
Partial clearance of warts at the end of treatment
Recurrence of any wart during the follow-up period
New warts during treatment and the follow-up period
Local sings and symptoms at the wart sites
Related adverse events during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Karl R. Beutner, M.D., Ph.D., Principal Investigator — Solano Clinical Research, 635 Anderson Road #17, Davis CA 95616, USA
Locations (12):
- United States (6):
  - Davis, San Diego, California
  - Denver, Colorado
  - New York, New York
  - Portland, Oregon
  - Houston, Dallas, Austin, Texas
  - Burlington, Vermont
- Buenos Aires, Argentina
- Santiago, Temuco, Chile
- Colombia, Bogota, Medellin, Risaralda, Colombia
- Cuautitlan, Mexico, Guadalajara, Durango, Ciliacan, Puebla, Mexico
- Lima, Calao, Peru
- Bucaresti, Brasov, Iasi, Cluj-Napoca, Romania

REFERENCES:
- [Derived] Tatti S, Swinehart JM, Thielert C, Tawfik H, Mescheder A, Beutner KR. Sinecatechins, a defined green tea extract, in the treatment of external anogenital warts: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1371-9. doi: 10.1097/AOG.0b013e3181719b60. PMID 18515521